CLINICAL TRIAL: NCT04632836
Title: Consequences of Respiratory Devices on Caregivers: CAP2 Study
Brief Title: Consequences of Respiratory Devices on Caregivers (CAP2)
Acronym: CAP2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asten Sante (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-ASTE-01; 20.06.11.64653 (Registry Identifier: SI CNRIPH number); 2020-A01741-38 (Other: ID RCB)
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Quality of Life
Keywords: quality of life; Home respiratory equipment; caregivers; Non-invasive ventilation; continuous positive airway pressure; long term oxygen therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NIV participant (non invasive-ventilation participant): From patient:
  * demographics data (date of birth, gender, socio-professional category, education level, morphometric data)
  * equipment data (type, indication, parameters, observance, usage data),
  * medical data (EFR, blood gas, respiratory polygraphy, pulse oxymetry, medical history, smoking status)
  * responses of questionnaires (WHOQOL-BREF questionnaire, PSQI index, HADS scale, study specific questionnaire)
  From partner:
  * demographics data (date of birth, gender, socio-professional category, education level, morphometric data)
  * responses of questionnaires (WHOQOL-BREF questionnaire, PSQI index, HADS scale, study specific questionnaire)
  Interventions: Other: quality of life questionnaires
- CPAP participant (continuous positive airway pressure participant): From patient:
  * demographics data (date of birth, gender, socio-professional category, education level, morphometric data)
  * equipment data (type, indication, parameters, observance, usage data),
  * medical data (EFR, blood gas, respiratory polygraphy, pulse oxymetry, medical history, smoking status)
  * responses of questionnaires (WHOQOL-BREF questionnaire, PSQI index, HADS scale, study specific questionnaire)
  From partner:
  * demographics data (date of birth, gender, socio-professional category, education level, morphometric data)
  * responses of questionnaires (WHOQOL-BREF questionnaire, PSQI index, HADS scale, study specific questionnaire)
  Interventions: Other: quality of life questionnaires
- LTOT participant (long term oxygen therapy participant): From patient:
  * demographics data (date of birth, gender, socio-professional category, education level, morphometric data)
  * equipment data (type, indication, parameters, observance, usage data),
  * medical data (EFR, blood gas, respiratory polygraphy, pulse oxymetry, medical history, smoking status)
  * responses of questionnaires (WHOQOL-BREF questionnaire, PSQI index, HADS scale, study specific questionnaire)
  From partner:
  * demographics data (date of birth, gender, socio-professional category, education level, morphometric data)
  * responses of questionnaires (WHOQOL-BREF questionnaire, PSQI index, HADS scale, study specific questionnaire)
  Interventions: Other: quality of life questionnaires

INTERVENTIONS:
Other: quality of life questionnaires — responses for quality of life questionnaires (WHOQOL-BREF questionnaire, study specific questionnaire, PSQI index, HADS scale)

SUMMARY:
The promoter of the study will conduct a monocentric cohort study that aim to evaluate the consequences of home respiratory devices on patient caregivers' quality of life.

The investigators will examine the impact of home respiratory devices on quality of life in general, sleep quality, anxiety and humour depending on equipment type (Non-invasive ventilation (NIV), continuous positive airway pressure (CPAP) or long-term oxygen therapy (LTOT)) for patients and partners. The investigators will assess the correlation between patient and caregiver's answers. The investigators will assess the correlation between couple's quality of life and adherence to treatment.

To do this, the investigators will use four quality of life questionnaires and the investigators will collect demographic data, medical data and usage report from the equipment.

DETAILED DESCRIPTION:
Home respiratory devices improve patients' quality of life and clinical outcomes. However, they bring medical equipment into the bedroom and are used overnight. The aim of this prospective cohort is to assess the quality of life of patient's caregivers.

Patient caregivers' quality of life will be assessed using the WHOQOL-BREF questionnaire (World Health Organization Quality of Life - Brief version questionnaire).

The investigators expect to enroll 200 patients' partners equipped with non-invasive ventilation, 100 patients' partners equipped with continuous positive airway pressure and 50 patients' partners equipped with long-term oxygen therapy. Patients will be recruited from the cohort of patients already established on home treatment and cared for by Asten Santé.

After consent, patient will receive dedicated questionnaires. During a home visit, home healthcare provider technician will retrieve data from the home device.

ELIGIBILITY:
Inclusion Criteria:

For the patient :

* Patient with a diagnostic of chronic obstructive pulmonary disease (COPD), sleep apnea or obesity hypoventilation syndrome
* Home respiratory equipment (NIV, CPAP or LTOT) since more than 3 months, patient and partner who shared the same household
* patient with medical stable condition
* patient who consents
* patient older than 18 years old
* patient followed at Rouen University Hospital

For the partner :

* patient who consents
* patient older than 18 years old

Exclusion Criteria:

For the patient :

* Home respiratory equipment for neuromuscular disease
* Patients who are institutionalized, deprived of their liberty or placed under judicial protection (guardianship or curatorship)
* patient not able to consent

For the partner :

* Patients who are institutionalized, deprived of their liberty or placed under judicial protection (guardianship or curatorship)
* patient not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Partners of adults patients who have home respiratory devices for chronic obstructive pulmonary disease (COPD), sleep apnea or obesity hypoventilation syndrome or other respiratory insuffisance disease and who share a same household.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Partner's quality of life score evaluated with WHOQOL-BREF questionnaire (World Health Organization Quality of Life - Brief version questionnaire) | The assessment will take place during the inclusion call (or in the following 10 days, during the respiratory devices provider's visit if the participant was unavailable to answer to the questionnaire during the inclusion call)
  Total quality of life score on WHOQOL-BREF questionnaire (World Health Organization Quality of Life - Brief version questionnaire). This questionnaire contains 26 items and addresses four quality of life domains. Items are rated on a 5-point Likert scale (low score of 1 to high score of 5) to determine a raw item score. The first and the second questions of the questionnaire are examined separately. For the other questions, the mean score for each domain is calculated, resulting in a mean score per domain that is between 4 and 20. Finally, this mean domain score is then multiplied by 4 in order to transform the domain score into a scaled score . For each domain, the minimum domain score is 4 and the maximum domain score is 20. It corresponds to a minimum scaled score of 0 and a maximum scale score of 100 for each domain. A higher score indicating a higher QOL.

SECONDARY OUTCOMES:
Partner's quality of life score evaluated with WHOQOL-BREF questionnaire (World Health Organization Quality of Life - Brief version questionnaire) for each equipment type | The assessment will take place during the inclusion call (or in the following 10 days, during the respiratory devices provider's visit if the participant was unavailable to answer to the questionnaire during the inclusion call)
  Total quality of life score on WHOQOL-BREF questionnaire (World Health Organization Quality of Life - Brief version questionnaire). This questionnaire contains 26 items and addresses four quality of life domains. Items are rated on a 5-point Likert scale (low score of 1 to high score of 5) to determine a raw item score. The first and the second questions of the questionnaire are examined separately. For the other questions, the mean score for each domain is calculated, resulting in a mean score per domain that is between 4 and 20. Finally, this mean domain score is then multiplied by 4 in order to transform the domain score into a scaled score . For each domain, the minimum domain score is 4 and the maximum domain score is 20. It corresponds to a minimum scaled score of 0 and a maximum scale score of 100 for each domain. A higher score indicating a higher QOL.
Patient's quality of life score evaluated with WHOQOL-BREF questionnaire (World Health Organization Quality of Life - Brief version questionnaire) for each equipment type | The assessment will take place during the inclusion call (or in the following 10 days, during the respiratory devices provider's visit if the participant was unavailable to answer to the questionnaire during the inclusion call)
  Total quality of life score on WHOQOL-BREF questionnaire (World Health Organization Quality of Life - Brief version questionnaire). This questionnaire contains 26 items and addresses four quality of life domains. Items are rated on a 5-point Likert scale (low score of 1 to high score of 5) to determine a raw item score. The first and the second questions of the questionnaire are examined separately. For the other questions, the mean score for each domain is calculated, resulting in a mean score per domain that is between 4 and 20. Finally, this mean domain score is then multiplied by 4 in order to transform the domain score into a scaled score . For each domain, the minimum domain score is 4 and the maximum domain score is 20. It corresponds to a minimum scaled score of 0 and a maximum scale score of 100 for each domain. A higher score indicating a higher QOL.
Partner's quality of life evaluated with study specific questionnaire for each equipment type | The assessment will take place during the inclusion call (or in the following 10 days, during the respiratory devices provider's visit if the participant was unavailable to answer to the questionnaire during the inclusion call)
  Total quality of life score on study specific questionnaire. It corresponds with the total score on the study specific questionnaire prepared by the investigators before the study after consulting a committee of experts in the field of chronic respiratory failure and a panel of patients familiar with ventilation according to the Delphi method. This questionnaire assesses five areas of quality of life : sleep, health, married life, social relations and participation in care through the 20 questions considered the most relevant by the panel.
  Items are rated on a 10-point Likert scale (low score of 0 to high score of 10) to determine each question score. For each question, the minimum score value is 0 and the maximum score value is 10. The minimum total score value is 0 reflection of a very negative impact of the equipment on the studied domains and the maximum score is 200, reflection of a very positive impact of the equipment.
Patient's quality of life evaluated with study specific questionnaire for each equipment type | The assessment will take place during the inclusion call (or in the following 10 days, during the respiratory devices provider's visit if the participant was unavailable to answer to the questionnaire during the inclusion call)
  Total quality of life score on study specific questionnaire. It corresponds with the total score on the study specific questionnaire prepared by the investigators before the study after consulting a committee of experts in the field of chronic respiratory failure and a panel of patients familiar with ventilation according to the Delphi method. This questionnaire assesses five areas of quality of life : sleep, health, married life, social relations and participation in care through the 20 questions considered the most relevant by the panel.
  Items are rated on a 10-point Likert scale (low score of 0 to high score of 10) to determine each question score. For each question, the minimum score value is 0 and the maximum score value is 10. The minimum total score value is 0 reflection of a very negative impact of the equipment on the studied domains and the maximum score is 200, reflection of a very positive impact of the equipment.
Partner's sleep quality evaluated with PSQI index (Pittsburgh Sleep Quality index) for each equipment | The assessment will take place during the inclusion call (or in the following 10 days, during the respiratory devices provider's visit if the participant was unavailable to answer to the questionnaire during the inclusion call)
  Total sleep quality score on PSQI index (Pittsburgh Sleep Quality index). The PSQI score will be expressed as a sub-score for the 7 areas of study and as an overall score (addition of all the sub-scores). For each studied domain, the minimum sub-score is 0 (best quality of sleep) and the maximum sub-score is 3 (worst quality of sleep). An overall score greater than or equal to 5 is a reflection of poor quality of sleep.
Patient's sleep quality evaluated with PSQI index (Pittsburgh Sleep Quality index) for each equipment | The assessment will take place during the inclusion call (or in the following 10 days, during the respiratory devices provider's visit if the participant was unavailable to answer to the questionnaire during the inclusion call)
  Total sleep quality score on PSQI index (Pittsburgh Sleep Quality index). The PSQI score will be expressed as a sub-score for the 7 areas of study and as an overall score (addition of all the sub-scores). For each studied domain, the minimum sub-score is 0 (best quality of sleep) and the maximum sub-score is 3 (worst quality of sleep). An overall score greater than or equal to 5 is a reflection of poor quality of sleep.
Partner's anxiety and humour score evaluated with HADS index (Hospital Anxiety and Depression scale) for each equipment | The assessment will take place during the inclusion call (or in the following 10 days, during the respiratory devices provider's visit if the participant was unavailable to answer to the questionnaire during the inclusion call)
  Total depression and anxiety score on HADS index (Hospital Anxiety and Depression scale). The HADS scale is an instrument used to screen for anxiety and depressive disorders. It has 14 items ranked from 0 to 3. Seven questions relate to anxiety and seven others to the depressive dimension. The score obtained on the HADS scale will be expressed as a score for each area of study:
  * the "anxiety score", evaluated by the 7 questions (questions number 1,3,5,7,9,11 and 13)
  * the depression score evaluated by the 7 other questions. The total score ranges from 0 to 42 for each participant. For each score (anxiety or depression), a score value of 7 or less corresponds to the absence of anxiety or depression. A score value between 8 and 10 reflects a doubtful symptomatology. A score value more than 11 reflect that the symptomatology is certain.
Patient's anxiety and humour score evaluated with HADS index (Hospital Anxiety and Depression scale) for each equipment | The assessment will take place during the inclusion call (or in the following 10 days, during the respiratory devices provider's visit if the participant was unavailable to answer to the questionnaire during the inclusion call)
  Total depression and anxiety score on HADS index (Hospital Anxiety and Depression scale). The HADS scale is an instrument used to screen for anxiety and depressive disorders. It has 14 items ranked from 0 to 3. Seven questions relate to anxiety and seven others to the depressive dimension. The score obtained on the HADS scale will be expressed as a score for each area of study:
  * the "anxiety score", evaluated by the 7 questions (questions number 1,3,5,7,9,11 and 13)
  * the depression score evaluated by the 7 other questions. The total score ranges from 0 to 42 for each participant. For each score (anxiety or depression), a score value of 7 or less corresponds to the absence of anxiety or depression. A score value between 8 and 10 reflects a doubtful symptomatology. A score value more than 11 reflect that the symptomatology is certain.
Correlation between patient's answers and partner's answers for each questionnaire | statistics through study completion, an average of 6 months
  Correlation between patient's answers and partner's answers for WHOQOL-bref questionnaire (World Health Organization Quality of Life - Brief version questionnaire) Correlation between patient's answers and partner's answers for study specific questionnaire Correlation between patient's answers and partner's answers for PSQI index (Pittsburgh Sleep Quality index) Correlation between patient's answers and partner's answers for HADS index (Hospital Anxiety and Depression scale)
Correlation between patient's answers and his observance | statistics through study completion, an average of 6 months
  Correlation between patient's answers for four questionnaires (World Health Organization Quality of Life - Brief version questionnaire, study specific questionnaire, Pittsburgh Sleep Quality index and Hospital Anxiety and Depression scale) and patient's observance data
Correlation between partner's answers and patient's observance | statistics through study completion, an average of 6 months
  Correlation between partner's answers for four questionnaires (World Health Organization Quality of Life - Brief version questionnaire, study specific questionnaire, Pittsburgh Sleep Quality index and Hospital Anxiety and Depression scale) and patient's observance data

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Patout, Principal Investigator — APHP-Sorbonne Université, Service des Pathologies du Sommeil (Département R3S) Paris, France
Locations (1):
- Asten Sante, Isneauville, France

IPD SHARING:
Plan to Share IPD: Yes
All specific individual participant data that underlie results in a publication will be made available upon reasonable request to the principal investigator
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available at the end of the study for time necessary to published and over a maximum of fifteen years (maximum time to store data on the online platform)
Access Criteria: Upon reasonable request to the principal investigator